CLINICAL TRIAL: NCT05111522
Title: Health-related Quality of Life (HRQoL) and Physical, Psychological and Cognitive Impairments After Intensive Care Unit (ICU)Discharge A Longitudinal Cohort Study
Brief Title: Health-related Quality of Life and Functional Impairments After Intensive Care Unit Discharge
Acronym: CritiQoL2
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Versailles Hospital (Other)
Collaborators: Legriel Stéphane (Unknown)
Responsible Party: Principal Investigator, Jacq Gwenaelle, principal investigator, Versailles Hospital
Other Study IDs: P21/07_CritiQol2
Record Dates: First submitted 2021-09-28; First posted 2021-11-08 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Health-related Quality of Life
Keywords: Health-related quality of life; Morbidity; Long terms outcomes; Post intensive care syndrome; Intensive Care Unit
MeSH Terms: conditions — postintensive care syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Diagnostic and therapeutic progress of the last twenty years has been accompanied by an evolution in the morbidity and mortality of intensive care unit (ICU) patients. While there has been an overall decrease in mortality in the ICU, nearly 20% of patients die within one year after ICU discharge and survivors are marked by an increase in morbidity.

Indeed, independently of the initial disease, it is currently recognized that an admission to the ICU can be experienced as a traumatic situation, with potential physical, psychological and cognitive impairments that can be described by the term "post-intensive care syndrome" (PICS). This results in a decrease in quality of life compared to the general population.

Health-related quality of life (HRQoL)has received increasing attention in the literature. Thus, many studies have been interested in its evaluation, in particular in certain pathologies such as acute respiratory distress syndrome (ARDS), sepsis, cardiac arrest or in patients with onco-hematological diseases.

Paradoxically, few studies have described the HRQoL and the elements of the PICS in the overall population of patients admitted to the ICU. However, a better understanding of these elements could allow us to propose improvement strategies to facilitate the rehabilitation of these patients.

DETAILED DESCRIPTION:
The investigators therefore propose the constitution of a longitudinal cohort evaluating the HRQoL, and allowing the analysis of its determinants in the global population of intensive care patients.

ELIGIBILITY:
Inclusion Criteria:

* all adult patients(age>18) hospitalized in ICU

Exclusion Criteria:

* legal guardianship
* opposition to participate
* unread and unwritten French language

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients who meet the eligibility criteria will be offered participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of an overall HRQOL and ii) percentage functional impairments in the global population of intensive care unit survivors,2 years after ICU discharge.according to the score to following scales : | 24month
  i)36-Item Short Form Survey (SF-36) (HRQoL)-Ranging score[0-100], a high score indicate better health status.
  ii)The Glasgow Outcome Scale extended (Handicap)-Ranging score[1-8] a hight score indicate no handicap.
  Barthel index (Dependency)-Ranging score[0-100], a high score indicate no dependency.
  The Fatigue Severity Scale(fatigue)-Ranging score[9-63],a high score indicate a greater fatigue severity.
  The Hospital anxiety and depression (Anxiety,Depression)-Ranging score[0-21] a score > 8 indicate in each subscale a depresion or/and anxiety The Impact of Event Scale -Revised(post traumatic syndrome disorder)-Ranging score[0-88],scores higher than 24 are of concern; the higher scores indicate the severity of PTSD The Montreal Cognitive Assessment (MoCA)(Cognition)-Ranging score[0-30] a score of 26 and higher generally is considered normal or Telephone MoCA-Ranging score[0-22],a score of 18 and higher generally is considered normal.

SECONDARY OUTCOMES:
Presence or not of elements associated with i) HRQOL impairements defined by ii)physical and/or psychological and /or cognitive impairments in the global population and in differents sub-groups of interest, according to the to following scales : | 24 month
  i)36-Item Short Form Survey (SF-36) (HRQoL)-Ranging score[0-100], a high score indicate better health status.
  ii)The Glasgow Outcome Scale extended (Handicap)-Ranging score[1-8] a hight score indicate no handicap.
  Barthel index (Dependency)-Ranging score[0-100], a high score indicate no dependency.
  The Fatigue Severity Scale(fatigue)-Ranging score[9-63],a high score indicate a greater fatigue severity.
  The Hospital anxiety and depression (Anxiety,Depression)-Ranging score[0-21] a score > 8 indicate in each subscale a depresion or/and anxiety The Impact of Event Scale-Revised(post traumatic syndrome disorder)-Ranging score[0-88],scores higher than 24 are of concern; the higher scores indicate the severity of PTSD The Montreal Cognitive Assessment (MoCA)(Cognition)-Ranging score[0-30] a score of 26 and higher generally is considered normal or Telephone MoCA-Ranging score[0-22],a score of 18 and higher generally is considered normal..

CONTACTS AND LOCATIONS:
Overall Officials: Gwenaëlle JACQ, RN,MSc, Principal Investigator — Versailles Hospital
Locations (1):
- Versailles hospital, Le Chesnay, France

IPD SHARING:
Plan to Share IPD: No